CLINICAL TRIAL: NCT00601146
Title: Low-Dose Chest Computed Tomography Screening for Lung Cancer in Survivors of Hodgkin's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Andrea K. Ng, MD, Radiation Oncologist, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 06-122
Record Dates: First submitted 2008-01-15; First posted 2008-01-25 (Estimated); Results first posted 2016-02-17 (Estimated); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Lung Cancer
Keywords: Hodgkin's disease; CT scan
MeSH Terms: conditions — Lung Neoplasms; Hodgkin Disease

STUDY DESIGN:
Intervention Model Description: Single arm study of low-dose Chest CT screening for long-term Hodgkin lymphoma survivors
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low-dose Chest CT screening (Experimental): Annual low-dose Chest CT screening
  Interventions: Procedure: chest computed tomography scan

INTERVENTIONS:
Procedure: chest computed tomography scan — Once a year for three years
  Other Names: CT scan

SUMMARY:
This research study is being done because patients with a history of chest radiation treatment for Hodgkin's disease have been shown to be at increased risk for developing lung cancer a number of years out from treatment. The risk appears to be further increased among patients with a smoking history. Currently, the practice is to recommend annual low-dose chest CT scans in survivors of Hodgkin's disease who have received prior chest radiation treatment and who have at least a moderate smoking history. In this study, the CT scans will be read and interpreted by the study radiologist, and the results recorded in a consistent manner.

DETAILED DESCRIPTION:
- Participants will undergo a chest computed tomography (CT) scan once a year for a 3-year period.

ELIGIBILITY:
Inclusion Criteria:

* 5 years or longer from initial Hodgkin's disease diagnosis
* Current age 18 or older
* Received mediastinal irradiation and/or alkylating-agent based chemotherapy
* Smoking history of 10-pack years or more, or current smoker
* Pre-approval from the participant's insurance company for the CT study

Exclusion Criteria:

* Patients with a history of lung cancer
* Currently receiving treatment for another cancer diagnosis
* Known diagnosis of any metastatic cancer
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2006-11-01; Primary Completion 2010-12-01 (Actual); Study Completion 2019-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea K. Ng, MD, Principal Investigator — Dana-Farber Cancer Institute/Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Low-dose CT Screening: Annual low-dose chest CT screening
Period: Overall Study
Arm/Group | Low-dose CT Screening
Started | 39
Completed (Study stopped early due to low accrual. Study is close to enrollment) | 39
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Low-dose CT Screening
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 51 [38 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: To Prospectively Collect Data on Chest CT Screening for Patients at Increase Lung-cancer Risk After Hodgkin's Disease.
Description: In this study, patients will under annual low-dose chest CT screening. The total number of lung cancer detected through the screening will be recorded
Time Frame: 3 years
Population: Enrolled patients who underwent low-dose CCT screening- number of lung cancer diagnosed
Measure: Number; unit: participants
Arm/Group | Low-dose CT Screening
Number analyzed (Participants) | 36
participants | 0

ADVERSE EVENTS:
Arm/Group | Low-dose CT Screening
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No